CLINICAL TRIAL: NCT06345820
Title: Intermediate Visual Acuity Comparison of Two Non-diffractive Enhanced Monofocal Intraocular Lenses
Brief Title: Comparison of Two Non-diffractive Enhanced Monofocal Intraocular Lenses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Evolux
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Cataract
Keywords: Cataract; Cataract surgery; Intraocular lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evolux (Experimental): Patient will receive the Enova IOL during cataract surgery
  Interventions: Device: Evolux
- Tecnis Eyhance (Experimental): Patient will receive the Tecnis Ehance IOL during cataract surgery
  Interventions: Device: Tecnis Eyhance

INTERVENTIONS:
Device: Evolux — Evolux, enhanced monofocal IOL
  Arms: Evolux
Device: Tecnis Eyhance — Tecnis Eyhance, enhanced monofocal IOL
  Arms: Tecnis Eyhance

SUMMARY:
Comparison of the clinical performance of two enhanced monofocal IOLs with similar design.

DETAILED DESCRIPTION:
In modern cataract surgery the aim of the procedure is not just the restoration of vision but to also achieve some spectacle independence. Bilateral implantation of monofocal intraocular lenses (IOL) aiming for emmetropia lead to high patient satisfaction levels in distance vision but leave patients dependent on spectacles in intermediate and near vision tasks.

To achieve high levels of spectacle independence the most commonly used option are multifocal intraocular lenses (MIOL). These MIOLs use either a refractive or diffractive optical design, a combination of both or segmented asymmetric optics. Usually, the characteristic diffractive ring patterns are incorporated on the posterior surface of an IOL, whereas the anterior lens surface remains purely refractive. However, a portion of patients experience problems with positive dysphotopsia symptoms such as halos and glare. Other potentially negative aspects of MIOLs are pupil size dependency and loss of light energy to higher order diffraction which can lead to reduced contrast sensitivity. In clinical studies diffractive lenses resulted in a better outcome in terms of optical quality, better contrast sensitivity and positive dysphotopsia phenomena than refractive multifocal lenses.

A newer concept of IOLs are non-diffractive enhanced range of vision (EROV) IOLs, sometimes also referred to as EDOF IOLs. The EROV IOLs with the least compromise concerning quality of vision are the group of so called enhanced monofocal IOL, also sometime referred to as monofocal plus IOL. These IOLs should result in better intermediate vison and provide contrast sensitivity and dysphotopsia results comparable to standard monofocal IOLs. These IOLs may be more adequate to meet the expectations of many presbyopic cataract patients, who were used to have a good distance vision and who were wearing spectacles when performing near vision tasks before surgery.

The aim of this study is to compare the clinical performance of a newer enhanced monofocal IOL (Evolux) with a standard enhanced monofocal IOL, the Tecnis Eyhance.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral cataract
* Age 21 or older
* Visual acuity > 0.05
* Axial length: 22.00-26.00mm
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Written informed consent prior to surgery
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures

Exclusion Criteria:

* Active ocular disease (e.g. chronic uveitis, proliferative diabetic retinopathy, chronic glaucoma not responsive to medication)
* Relevant other ophthalmic diseases such as pseudoexfoliation syndrome (PEX), Intraoperative Floppy Iris Syndrome (IFIS)
* Corneal decompensation or corneal endothelial cell insufficiency
* Amblyopia
* Previous ocular surgery or trauma
* Persons who are pregnant or nursing (pregnancy test will be taken in women of reproductive age)
* Astigmatism with the need for a toric IOL

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Monocular intermediate visual acuity | 24 months
  Monocular intermediate visual acuity at 66 cm will be measured using ETDRS charts

SECONDARY OUTCOMES:
Monocular distance visual acuity | 24 months
  Monocular distance visual acuity at 4 meters will be measured using ETDRS charts
Monocular near visual acuity | 24 months
  Monocular near visual acuity at 40 cm will be measured using ETDRS charts

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Prim. Dr., Principal Investigator — Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Krankenhaus
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided